CLINICAL TRIAL: NCT03146754
Title: A Study to Evaluate Lung Ultrasound as a Method to Measure Changes in Extravascular Lung Water Induced by Positional Changes or Exercise in Patients Stabilized Following Hospitalization for Acute Decompensated Heart Failure
Brief Title: A Study to Evaluate Lung Ultrasound as a Method to Measure Changes in Extravascular Lung Water Induced by Positional Changes (LUPE)
Acronym: LUPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 827232
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Acute Decompensated Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stable ADHF patients (Experimental): Lung ultrasound to access b lines
  Interventions: Other: Methodology
- Control Patients (Active Comparator): Patients without any cardiopulmonary disease will be control patients for the active subjects, age-matched accordingly.
  Interventions: Other: Methodology

INTERVENTIONS:
Other: Methodology — No intervention will be performed. Study is designed to test methodology of lung ultrasound in accessing b lines (2 phases)

SUMMARY:
This is an exploratory study to evaluate lung ultrasound as a method for measuring extravascular lung water in stabilized patients during hospitalization for ADHF. Subjects who have been stabilized following admission for ADHF and capable of lying supine will be evaluated by lung ultrasound to determine the degree of lung congestion as measured by the total B-line score. Since different patients may require different degrees of postural change and/or other maneuvers (e.g., leg elevation or exercise) to induce B-line increments, a tailored sequential protocol will be employed to define which maneuvers are sufficient for each patient. Control patients, age-matched, will be recruited to provide a comparison group for data analysis.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized for the management of acute decompensated heart failure

Reached at least a 12-hour period after hospital admission

Presence of peripheral edema with a score of at least 1+ (slight pitting in both ankles; 2mm or less depression that disappears rapidly)

Able to lie supine with no more than one pillow (approximately a 10 cm head elevation) without dyspnea for at least 30 minutes by patient report

Have not received treatment with any intravenous loop diuretic within the 4 hours prior to initiating study assessments and with no plans for additional intravenous treatment during the series of lung ultrasound measurements

Exclusion Criteria:

Persistent uncontrolled hypertension (resting systolic blood pressure > 160 mmHg)

Significant lung disease including severe chronic obstructive pulmonary disease (See concomitant medication exclusions), pulmonary fibrosis, active asthma or acute pneumonia

Use of medications specified for the treatment of COPD including short- and long-acting bronchodilators (β-agonists and anticholinergics) and inhaled glucocorticoids as well as oxygen therapy

Use of another investigational product in a clinical study within the following time period prior to the first administration of study medication: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change in B-line score | Day 1
  Measured by lung ultrasound
Change in B-line score | Day 1
  Change in B-line score with leg elevation (in those subjects undergoing assessment)
Change in B-line score | Day 1
  Change in B-line score with the transition to a Trendelenberg position where the head is 10 degrees lower than the feet (in those subjects undergoing assessment)
Change in B-line score | Day 1
  Change in B-line score with exercise (in those subjects undergoing assessment)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De identified IPD will be shared with collaborators